CLINICAL TRIAL: NCT06479434
Title: Association of Serum Biomarkers in Polycystic Ovarian Syndrome (PCOS) Females With and Without Metformin Versus Healthy Controls
Brief Title: Serum Biomarker Levels Improvement in Poly Cystic Ovarian Syndrome: Impact of Metformin Compared to Healthy Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: University of Karachi (Other)
Responsible Party: Principal Investigator, Sadia Fatima, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 08232/SC
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2024-06

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin Treated PCO (Experimental): After taking informed consent demographic data like name, age, anthropometric measurements (blood pressure, BMI, weight, height)will be recorded by researcher Body mass index (BMI), waist circumference, waist to hip ratio will be evaluated. Blood samples will be collected after an overnight fast of 8 to 10 hours. Then metformin will be given to subjects a dose of 500 mg three times a day for 8 weeks. Serum biomarkers and inflammatory markers will be assessed at day 0 and after 8 weeks post metformin administration.
  Interventions: Drug: Metformin
- PCO without Metformin (No Intervention): After taking informed consent demographic data like name, age, anthropometric measurements (blood pressure, BMI, weight, height)will be recorded by researcher Body mass index (BMI), waist circumference, waist to hip ratio will be evaluated. Blood samples will be collected after an overnight fast of 8 to 10 hours. . Serum biomarkers and inflammatory markers will be assessed at day 0 only.

INTERVENTIONS:
Drug: Metformin — Females diagnosed with polycystic syndrome will be given metformin tablets for 8 weeks and followed up. Blood samples will be collected along with anthropometric data (weight (kg), height (m) etc)
  Arms: Metformin Treated PCO

SUMMARY:
The goal of this interventional study is to assess the effect of drug metformin in improving the fertility hormones and reducing the inflammatory hormones in polycystic ovarian syndrome (PCOS) patients. We wish to answer the question whether metformin is necessary to improve PCOS symptoms versus simple lifestyle modification.

Participants once diagnosed with PCOS will be given metformin to be sued for 8 weeks. They will be asked to provide blood samples on day 0 and after 8 weeks of metformin use. The blood sample will be used to measure the hormonal and inflammatory profile. In addition, they will be required to compete a questionnaire regarding symptoms such as decrease in facial hair growth, improvement in menstrual cycle etc.

ELIGIBILITY:
Inclusion Criteria:

a) Patients Falling into PCOS as per Rotterdam criteria

Exclusion Criteria:

1. Systemic diseases like atherosclerosis,
2. Diabetes mellitus
3. Hypertension
4. congenital adrenal hyperplasia, androgen secreting tumors

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Change in hormonal profile and menstural Cycle after Metformin use | 8 weeks
  Serum reproductory hormone levels (follicle stimulating hormone, testosterone), inflammatory hormones (tumor necrosis factor, c reactive protein) will be measured at day 0 and after 8 weeks of intervention

SECONDARY OUTCOMES:
Change in symptoms associated with PCO after intervention | 8 weeks
  Subjects will be asked to score on a Likert scare (0-5) change in the mood swings, menstural cycle frequency, facial hair quantity and quality, and dietary and bowel movement improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Sadia Fatima, PhD, Study Director — Aga Khan University
Locations (1):
- DBBS, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No